CLINICAL TRIAL: NCT06776770
Title: A Phase Ib/II Study of Adebrelimab in Combination with Capecitabine and Oxaliplatin in Previously Untreated Advanced or Metastatic Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Phase Ib/II Study of Adebrelimab in Combination with Capecitabine and Oxaliplatin in Cancer
Acronym: GC-Ib/II
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADE-GC-Ib/II-XELOX
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: Adebrelimab plus capecitabine and oxaliplatin
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab plus capecitabine and oxaliplatin (Experimental): Phase I: Cohort 1: Adebrelimab 10 mg/kg Q3W plus capecitabine and oxaliplatin (XELOX regimen); 21-day treatment cycle; Cohort 2: Adebrelimab 1200 mg or 20 mg/kg Q3W plus capecitabine and oxaliplatin (XELOX regimen); 21-day treatment cycle.
  Phase II: Adebrelimab (RP2D, Q3W) + (XELOX regimen), with a 3-week (21-day) treatment cycle.
  XELOX regimen：Oxaliplatin 130 mg/m2 iv.gtt d1，Capecitabine 1,000 mg/m2 p.o.b.i.d.d1~14
  Interventions: Drug: Adebrelimab

INTERVENTIONS:
Drug: Adebrelimab — Phase I: Cohort 1: Adebrelimab 10 mg/kg Q3W plus capecitabine and oxaliplatin (XELOX regimen); 21-day treatment cycle; Cohort 2: Adebrelimab 1200 mg or 20 mg/kg Q3W plus capecitabine and oxaliplatin (XELOX regimen); 21-day treatment cycle.
  Phase II: Adebrelimab (RP2D, Q3W) + (XELOX regimen), with a 3-week (21-day) treatment cycle.
  XELOX regimen：Oxaliplatin 130 mg/m2 iv.gtt d1，Capecitabine 1,000 mg/m2 p.o.b.i.d.d1~14.
  Other Names: Adebrelimab Injection

SUMMARY:
In this study, the combination of Adebrelimab (PD-L1 monoclonal antibody) on the basis of standard treatment (two-drug chemotherapy regimen of fluorouracil and platinum drugs) may enhance the immune response in order to enhance the killing effect on tumor cells and bring survival benefits to patients with advanced or metastatic gastric cancer or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
This study is divided into two phases: Phase Ib is a study on the tolerance and safety of Adebrelimab combined with capecitabine and oxaliplatin in the treatment of patients with advanced solid tumors; Phase II is a single-arm, open-label clinical study to observe and evaluate the improvement of objective response rate (ORR) in advanced or metastatic gastric cancer or gastroesophageal junction adenocarcinoma treated with adebrelimab combination therapy. A total of 52 subjects are expected to be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

- 1. The patients voluntarily participated in the study and signed the informed consent; 2. ≥ 18 years old (calculated on the day of signing informed consent), both male and female; 3. Patients with pathologically confirmed gastric cancer (GC) or gastroesophageal junction cancer (GEJC) who were histologically confirmed to be adenocarcinoma and had not received antineoplastic therapy for GC or GEJC; 4. No prior systemic therapy for advanced or metastatic disease. Prior adjuvant or neoadjuvant chemotherapy for GC and GEJC,Radiotherapy or chemoradiotherapy, provided that the last dose of the last drug (based on the last dose) occurred at least 6 months prior to enrollment. Palliative radiotherapy is allowed, but it must be completed 2 weeks before enrollment; 5. Human epidermal growth factor receptor 2 negative or unknown; 6. At least one measurable lesion according to the solid tumor efficacy evaluation criteria (RECIST v1.1); 7. The Eastern Cooperative Oncology Group (ECOG) physical status score was 0-1. 8. Expected survival > 12 weeks; 9. Adequate organ and bone marrow function, as defined below: A) Neutrophil count (ANC) ≥ 1,500/mm3 (1.5 × 10 ^ 9/L); B) Platelet count (PLT) ≥ 75,000/mm3 (75 × 10 ^ 9/L); C) hemoglobin (Hb) ≥ 8 G/dL (80 G/L); D) Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 40 ml/min; E) Total bilirubin (BIL) ≤ 1.5 times the upper limit of normal (ULN); F) Aspartate transaminase or Alanine transaminase ≤ 2.5 times the upper limit of normal (ULN), and ≤ 5 × ULN for patients with liver metastasis; G) International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN; H) Urine protein < 2 +; if urine protein ≥ 2 +, 24-hour urine protein quantification shows that protein must be ≤ 1 G; I) Thyroid-stimulating hormone (TSH) ≤ upper limit of normal (ULN); if abnormal, T3 and T4 levels should be investigated, and normal T3 and T4 levels can be included.

10.Female subjects of childbearing age must have a negative serum pregnancy test within 3 days prior to the start of study medication and be willing to use a medically approved highly effective contraceptive method (e.g., intrauterine device, contraceptive pill, or condom) for the duration of the study and for 3 months after the last dose of study medication; Male subjects with a female partner of childbearing age were surgically sterilized or agreed to use an effective method of contraception for the duration of the study and for 3 months after the last study dose.

Exclusion Criteria:

* 1. Previous treatment with PD-1/PD-L1 antibodies, cytotoxic T lymphocyte-associated antigen-4 antibodies, or other PD-1/PD-L1 inhibitors; 2. Past hypersensitivity to monoclonal antibodies and inactive ingredients of this product; 3. Previous use of immunosuppressive drugs within 14 days prior to the first dose of study drug, excluding nasal and inhaled corticosteroids or physiologic doses of systemic steroid hormones (i.e., up to 10 mg/day of prednisolone or pharmacophysiologically equivalent doses of other corticosteroids).； 4. Vaccination with live attenuated vaccine within 4 weeks before the first dose or planned during the study; 5. Patients with clinical signs and symptoms of central nervous system metastasis or other evidence that central nervous system metastasis has not been controlled are not suitable for inclusion according to the judgment of the investigator, and those with meningeal metastasis history or symptoms and signs need to be excluded; 6. Toxicity of previous antineoplastic therapy did not recover to the level of CTCAE v5.0 ≤ 1 or the level specified in the inclusion/exclusion criteria; except for other toxicities such as alopecia, which the investigator considered did not pose a safety risk to the patient; 7. Advanced patients with symptoms, dissemination to the viscera, and risk of life-threatening complications in the short term (including patients with uncontrollable massive exudates [thoracic, pericardial, abdominal], pulmonary lymphangitis, and liver involvement of more than 30%); 8. Presence of any active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis,Hyperthyroidism, hypothyroidism; subjects with vitiligo or complete remission of asthma in childhood without any intervention in adulthood can be included; subjects with asthma requiring medical intervention of bronchodilators can not be included); 9. Any other malignancy diagnosed within 3 years prior to study entry, except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix; 10. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive, and hepatitis C virus-RNA above the detection limit of the analytical method), or co-infection with hepatitis B and hepatitis C; 11.Myocardial infarction, severe/unstable angina, NYHA class 2 or greater cardiac dysfunction, and poorly controlled arrhythmias (including Corrected QT Interval interval > 450 ms in men and > 470 ms in women) within 6 months prior to study entry. QTcF interval was calculated by Fridericia formula), symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism); 12.Hypertension that is not well controlled by antihypertensive medication (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg); 13. Coagulation dysfunction (INR > 1.5 or APTT > 1.5 × ULN), bleeding tendency or receiving thrombolytic or anticoagulant therapy; 14. Known hereditary or acquired bleeding and thrombotic tendencies, such as hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc; 15. Patients with obvious hemoptysis or daily hemoptysis volume of half a teaspoon (2.5 ml) or more within 2 months before entering the study; 16. There were clinically significant bleeding symptoms or definite bleeding tendency within 3 months before entering the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood + + and above, or vasculitis; 17. Arterial/venous thrombotic events occurred within 6 months before entering the study, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism.

  18. Known hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.); 19. Long-term anticoagulation therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day); 20. Complicated with severe infection within 4 weeks before the first medication (e.g., need for intravenous antibiotics, antifungal or antiviral drug), or unexplained fever > 38.5 ° C during screening/before first dose; 21. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 22. Participated in any other clinical study of the drug within 4 weeks prior to the first dose, or not more than 5 half-lives from the last study dose; 23. Known history of psychotropic substance abuse or drug use; 24. Patients with other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study or interfere with the results of the study, and who are not considered suitable for participation in the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | 48 months
  Dose-limiting toxicity
Maximum tolerated dose (MTD) | 48 months
  Maximum tolerated dose
Recommended Dose for Phase II Clinical Study (RP2D) | 48 months
  Recommended Dose for Phase II Clinical Study
Objective Response Rate (ORR) | 48 months
  Objective Response Rate

SECONDARY OUTCOMES:
Median progression-free survival (PFS) | 48 months
  Median progression-free survival
Time-To-Progression (TTP) | 48 months
  Time-To-Progression
Disease control rate (DCR) | 48 months
  Disease control rate
Duration of Response (DoR) | 48 months
  Duration of Response
overall survival (OS) | 48 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Hospital, Cancer Hospital, Chinese Academy of Medical Sciences, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided